CLINICAL TRIAL: NCT05564819
Title: Efficacy and Safety of Acetaminophen in Postoperative Pain Management of Infants Under Enhanced Recovery After Surgery
Brief Title: Efficacy and Safety of Acetaminophen in Postoperative Pain Management of Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Weibing Tang, Chief of Department of neonatal surgery, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCH202207156
Record Dates: First submitted 2022-09-16; First posted 2022-10-04 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Analgesic; Enhanced Recovery After Surgery; Postoperative Pain; Infant ALL; Acetaminophen
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): After recovering and returning to the ward, acetaminophen (10mg/kg) was taken orally immediately; once every 6 hours, a total of 4 times.
  Interventions: Drug: Acetaminophen
- placebo group (Placebo Comparator): The same amount of sterilized water was administered orally at the same time points.
  Interventions: Drug: Sterilized water

INTERVENTIONS:
Drug: Acetaminophen — When the infants woke up after surgery and were transported back to the ward, they were randomly divided into two groups immediately. The intervention group was given oral acetaminophen, once every 6 hours, for a total of 4 times.
  Arms: Treatment group
Drug: Sterilized water — When the infants woke up after surgery and were transported back to the ward, they were randomly divided into two groups immediately. The control group was given sterilized water, once every 6 hours, for a total of 4 times.
  Arms: placebo group

SUMMARY:
Pain will bring early and long-term adverse reactions to infants. The investigators need to pay attention to whether there is pain in infants after surgery. Since infants cannot self-report pain,The investigators need to use appropriate pain assessment scale to evaluate the pain of these infants, so as to understand the status of postoperative pain in children. The result of pain score not only enables investigators to understand the pain status of children, but also helps investigators to give corresponding intervention and treatment according to the pain degree of children. Postoperative pain management is one of the core contents of ERAS. Effective pain management is beneficial to the early postoperative recovery of infants and reduces the adverse reactions caused by pain. Sveral studies have confirmed that the combination of acetaminophen and opioids could reduce the use of opioids after surgery. But even if opioid use is reduced, it still causes many side effects for children. This study evaluated the safety and efficacy of acetaminophen alone for postoperative analgesia in infants.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent was obtained from parents of children;
* Infants aged 0-12 months;
* Children who underwent abdominal and perineal surgery in the Department of Neonatal Surgery, Children's Hospital Affiliated to Nanjing Medical University and returned to the unaccompanied ward after removal of tracheal intubation.

Exclusion Criteria:

* No informed consent was obtained from parents;
* known allergy or intolerance to acetaminophen;
* Children with liver function impairment (alanine aminotransferase/aspartate aminotransferase (ALAT/ASAT) more than three times the reference value;
* Children with renal insufficiency (urea and creatinine values exceeding the upper limit of reference values);

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Using CRIES scale to assess the pain level at 12 hours after postoperative awakening | 12 hours after postoperative awakening
  The pain score was evaluated 12 hours after Children wake up

SECONDARY OUTCOMES:
liver function | 48 hours after surgery
  alanine aminotransferase, aspartate aminotransferase
renal function | 48 hours after surgery
  urea and creatinine values
LOS | 30 days after surgery
  Length of stay after surgery
Using CRIES scale to assess the pain level at 1 hour after postoperative awakening | 1 hour after postoperative awakening
  The pain score was evaluated 1 hour after Children wake up
Using CRIES scale to assess the pain level at 6 hours after postoperative awakening | 6 hours after postoperative awakening
  The pain score was evaluated 6 hours after Children wake up
Using CRIES scale to assess the pain level at 18 hours after postoperative awakening | 18 hours after postoperative awakening
  The pain score was evaluated 18 hours after Children wake up
Using CRIES scale to assess the pain level at 24 hours after postoperative awakening | 24 hours after postoperative awakening
  The pain score was evaluated 24 hours after Children wake up
Using CRIES scale to assess the pain level at 36 hours after postoperative awakening | 36 hours after postoperative awakening
  The pain score was evaluated 36 hours after Children wake up
Using CRIES scale to assess the pain level at 48 hours after postoperative awakening | 48 hours after postoperative awakening
  The pain score was evaluated 48 hours after Children wake up
Using FLACC scale to assess the pain level at 1 hour after postoperative awakening | 1 hour after postoperative awakening
  The pain score was evaluated 1 hour after Children wake up
Using FLACC scale to assess the pain level at 6 hours after postoperative awakening | 6 hours after postoperative awakening
  The pain score was evaluated 6 hours after Children wake up
Using FLACC scale to assess the pain level at 12 hours after postoperative awakening | 12 hours after postoperative awakening
  The pain score was evaluated 12 hours after Children wake up
Using FLACC scale to assess the pain level at 18 hours after postoperative awakening | 18 hours after postoperative awakening
  The pain score was evaluated 18 hours after Children wake up
Using FLACC scale to assess the pain level at 24 hours after postoperative awakening | 24 hours after postoperative awakening
  The pain score was evaluated 24 hours after Children wake up
Using FLACC scale to assess the pain level at 36 hours after postoperative awakening | 36 hours after postoperative awakening
  The pain score was evaluated 36 hours after Children wake up
Using FLACC scale to assess the pain level at 48 hours after postoperative awakening | 48 hours after postoperative awakening
  The pain score was evaluated 48 hours after Children wake up
Using CHIPPS scale to assess the pain level at 1 hour after postoperative awakening | 1 hour after postoperative awakening
  The pain score was evaluated 1 hour after Children wake up
Using CHIPPS scale to assess the pain level at 6 hours after postoperative awakening | 6 hours after postoperative awakening
  The pain score was evaluated 6 hours after Children wake up
Using CHIPPS scale to assess the pain level at 12 hours after postoperative awakening | 12 hours after postoperative awakening
  The pain score was evaluated 12 hours after Children wake up
Using CHIPPS scale to assess the pain level at 18 hours after postoperative awakening | 18 hours after postoperative awakening
  The pain score was evaluated 18 hours after Children wake up
Using CHIPPS scale to assess the pain level at 24 hours after postoperative awakening | 24 hours after postoperative awakening
  The pain score was evaluated 24 hours after Children wake up
Using CHIPPS scale to assess the pain level at 36 hours after postoperative awakening | 36 hours after postoperative awakening
  The pain score was evaluated 36 hours after Children wake up
Using CHIPPS scale to assess the pain level at 48 hours after postoperative awakening | 48 hours after postoperative awakening
  The pain score was evaluated 48 hours after Children wake up

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shi C, Tang J, Sun W, Li W, Lv X, Tang W. Efficacy and safety of oral paracetamol for the management of acute postoperative pain in neonates and infants: a randomized clinical trial. World J Pediatr Surg. 2026 Feb 3;9(1):e001131. doi: 10.1136/wjps-2025-001131. eCollection 2026. PMID 41657425